CLINICAL TRIAL: NCT03290703
Title: A Phase I, Single Center, Randomized, Open-Label Study Investigating the Effect of Formulation, Food, and Rabeprazole on the Pharmacokinetics of GDC-0853 in Healthy Subjects
Brief Title: A Study to Investigate the Effect of Formulation, Food, and Rabeprazole on the Pharmacokinetics (PK) of GDC-0853 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GP39619; 2017-000752-26 (EudraCT Number)
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — fenebrutinib; Rabeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: GDC-0853 (Effect of Formulation) (Experimental): Participants will receive five single oral doses of test formulations of GDC-0853 co-administered with rabeprazole in the fasted state.
  Interventions: Drug: GDC-0853; Drug: Rabeprazole
- Part 2: GDC-0853 (Effect of Food and Rabeprazole) (Experimental): Participants will receive three single oral doses of one GDC-0853 formulations selected from Part 1 of this study. One dose will be administered in the fasted state, one dose will be administered in the fed state, and one dose will be co-administered with rabeprazole in the fed or fasted state, depending on randomization.
  Interventions: Drug: GDC-0853; Drug: Rabeprazole
- Part 3: GDC-0853 Optimized (Effect of Food and Rabeprazole) (Experimental): Participants will receive three single oral doses of an optimized tablet formulations of GDC-0853. One dose will be administered in the fasted state, one dose will be administered in the fed state, and one dose will be co-administered with rabeprazole in the fed or fasted state, depending on randomization.
  Interventions: Drug: GDC-0853; Drug: Rabeprazole

INTERVENTIONS:
Drug: GDC-0853 — Participants will receive different formulations of GDC-0853 tablet.
  Other Names: RO7010939
Drug: Rabeprazole — Participants will receive rabeprazole 20 mg twice daily (BID) for three days prior to GDC-0853 administration and a single dose coadministered with GDC-0853.

SUMMARY:
The purpose of this study is to evaluate the PK of GDC-0853 following changes to formulation and in the presence or absence of food, the proton pump inhibitor (rabeprazole), or both. This will be a 3-part open-label randomized study conducted in healthy adult participants. Approximately 63 subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female (of non-childbearing potential) participants
* Within body mass index range 18.0 to 32.0 kilogram per meter square (kg/m^2), inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), vital signs and physical examinations
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* History or symptoms of any significant disease
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection
* Participants who previously participated in any other investigational study drug trial within 90 days prior to Check-in. Participants who previously received GDC-0853 in previous studies.
* History of malignancy
* Pregnancy, lactation, or breastfeeding in female participants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of GDC-0853 | Pre-dose (within 1 hour) and 0.5 hours up to 72 hours post-dose on Day 1 of each Part
Time to Reach Maximum Observed Plasma Concentration (Tmax) of GDC-0853 | Pre-dose (within 1 hour) and 0.5 hours up to 72 hours post-dose on Day 1 of each Part
Area Under the Curve From Time Zero to Last Measurable Concentration [AUC (0-t)] of GDC-0853 | Pre-dose (within 1 hour) and 0.5 hours up to 72 hours post-dose on Day 1 of each Part
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-inf)] of GDC-0853 | Pre-dose (within 1 hour) and 0.5 hours up to 72 hours post-dose on Day 1 of each Part
Extrapolated Area Under the Curve (AUC Percent [%] Extrap) of GDC-0853 | Pre-dose (within 1 hour) and 0.5 hours up to 72 hours post-dose on Day 1 of each Part
Apparent Terminal Elimination Rate Constant of GDC-0853 | Pre-dose (within 1 hour) and 0.5 hours up to 72 hours post-dose on Day 1 of each Part
Apparent Volume of Distribution (Vz/F) of GDC-0853 | Pre-dose (within 1 hour) and 0.5 hours up to 72 hours post-dose on Day 1 of each Part
Apparent Oral Clearance (CL/F) of GDC-0853 | Pre-dose (within 1 hour) and 0.5 hours up to 72 hours post-dose on Day 1 of each Part
Relative Bioavailability (Frel) of GDC-0853 | Pre-dose (within 1 hour) and 0.5 hours up to 72 hours post-dose on Day 1 of each Part
Apparent Terminal Elimination Half-Life (t1/2) of GDC-0853 | Pre-dose (within 1 hour) and 0.5 hours up to 72 hours post-dose on Day 1 of each Part

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | From screening to the end of the study (approximately a maximum of 11 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial, Study Director — Hoffmann-La Roche
Locations (1):
- Quotient Clinical Ltd, Clinical Research Unit, Nottingham, United Kingdom